CLINICAL TRIAL: NCT06690372
Title: Improving Cardiometabolic Health in Individuals With SCI Using Home-Based Interactive Virtual Gaming
Brief Title: Improving Heart Health in Individuals With SCI Using Home-Based Virtual Gaming
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Margaret A. Finley, Associate Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC230078CTA_VirtualReality; HT94252410878 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: spinal cord injury; cardiometabolic risk; virtual reality exercise; physical activity
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: A repeated measures, single group, crossover design will be used, with 16 participants. Once enrolled, participants will serve as their own control with a 4-week control phase (baseline) followed by participation in the 12-week home-based VR-Move exercise protocol (intervention phase).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preliminary clinical efficacy and feasibility of 12-week home-based VR-Move exercise program (Experimental): Following baseline (week 0) assessments participants will be instructed to maintain their daily activities as usual for four weeks. Following the 4-week control phase, and the pre-intervention data collection session participants will be provided with instructions on set-up and use of the VR exercise platform, clinical dashboard and mobile app. Participants will be issued a wireless heart rate monitor (Polar Electro Oy, Model 190027141, Kemple, Finland) to wear on their wrist during each exercise session, tracking heart rate. Participants will be asked to use the VR-Move platform independently following system prompts (as with any virtual exercise product). Over the 12-weeks, participants will be instructed to exercise with the VR-Move 3x/week for 30 minutes for 12-weeks total, with modules presented in a prescribed weekly sequence to provide novel and re-enforcement of modules, while ensuring all modules are performed. Further, participants will be provided the opportunity of a 30 m
  Interventions: Other: virtual reality exercise

INTERVENTIONS:
Other: virtual reality exercise — Over the 12-weeks, participants will be instructed to exercise with the VR-Move 3x/week for 30 minutes for 12-weeks total, with modules presented in a prescribed weekly sequence to provide novel and re-enforcement of modules, while ensuring all modules are performed. Further, participants will be provided the opportunity of a 30 minute "free-play" of module of choice once a module has been introduced.

SUMMARY:
What is the ultimate applicability of the research? Individuals with SCI face several challenges when trying to engage in exercise following injury. Barriers to engagement include cost, transportation, and lack of SCI accessible resources. At the same time, individuals with SCI are at risk of developing negative health consequences (e.g., cardiovascular disease) associated with physical inactivity. A critical need exists to improve relevant, accessible, and sustainable home-based exercise interventions for individuals with SCI to lower the risk of developing secondary comorbid diseases from physical inactivity and to promote wellness. This research will investigate a fun and novel in-home virtual reality system aimed toward improving physical fitness of individuals SCI with the ultimate goal of improving physical, emotional, and psychosocial quality of life. Virtual reality gaming has been used for a long time to improve physical fitness, but there have yet to be virtual reality games designed specifically for individuals with SCI. The explicit aim of this research is therefore to develop a therapeutic technology that will be widely accessible to individuals with SCI.

What persons with SCI and/or their caregivers will it help, and how will it help them? We aim to provide a readily available exercise platform for individuals with SCI, across a spectrum of physical function. Research has shown that individuals with SCI are particularly prone to be physically inactive. The consequences of physical inactivity have been well documented and include negative outcomes in physical, psychological, and social health with reduced quality of life. For the current study, we will refine our existing virtual reality exercise platform, VR-Move with a focus on non ambulatory individuals with bilaterally preserved C6 function. Our focus on using the exercise platform for this cohort of the SCI population is meant to provide a basis for developing and catering to the platform for higher levels of SCI injury (higher quadriplegic). From our previous work with virtual reality interventions in SCI, we recognize that this product can be widely used by individuals across the age spectrum independently of their home environment.

What are the potential clinical applications, benefits, and risks? The proposed virtual reality exercise platform, VR-Move, is intended to provide one of the few accessible exercise modalities designed specifically for individuals with SCI and is readily adaptable across the clinical spectrum - including clinic and self-guided home use. There are no known risks associated with this research.

How will the pilot clinical trial advance the research findings along the translational spectrum? This project aims to refine and assess timely therapeutic technology with the specific intention of translating study findings into a clinically validated, widely accessible health product that can be deployed and implemented within the home. The project likewise demonstrates collaboration between academia, industry (a veteran-owned business), and veteran SCI communities. Project completion will offer initial validation of a novel health promoting modality (i.e., virtual reality exercise) informed by individuals living with SCI and experts in SCI to be relevant and responsive to specific health/exercise needs of persons living with SCI. Larger clinical trial testing will subsequently inform product commercialization and dissemination. The resulting platform, developed for unattended in-home use, is expected to make a meaningful contribution to SCI health and physical fitness, accessibility, and quality of life.

What is the projected time it may take to achieve a person-related outcome? The team is purposefully refining the existing exercise platform, VR-Move, so that it can be easily implemented within people's homes or in clinic settings. Pending findings from the pilot clinical study, this exercise platform would be available immediately to individuals with SCI

What are the likely contributions of the proposed research project to advancing the field of SCI research, patient care, and/or quality of life? The proposed study may make significant contributions across several areas. First, it will facilitate fruitful clinical data and basic lines of scientific inquiry regarding the application of the physical activity paradigm. The study will also increase our knowledge regarding the importance of consumer advocate-driven research for individuals with SCI. Second, low-activity following SCI is consistently associated with reduced quality of life among individuals with SCI and their families; access to an inexpensive portable intervention will therefore significantly improve quality of life among those affected by low-activity SCI.

DETAILED DESCRIPTION:
Overview. Cardiovascular diseases (coronary heart disease, myocardial infarction, stroke) have emerged as leading sources of illness and death for persons with spinal cord injury (SCI). Cardiometabolic disease/syndrome (CMD) is a central risk factor for both cardiovascular disease and diabetes mellitus, and encompasses a cluster of risk factors including hypertension, dyslipidemia, elevated glucose profiles, and central adiposity. In comparison to the general populations, individuals with SCI are more likely to develop CVD and are more likely to have cardiovascular disease and diabetes mellitus. The prevalence of CMD in the SCI population ranges from 33%5 and 63%, and one study found that nearly 58% of Veterans with SCI presented with CMD. Physical inactivity is associated with multiple components of CMD, including obesity, insulin resistance, hypertension, and dyslipidemia. However, while moderate intensity exercise is supported as a powerful tool against CMD over half of individuals living with SCI report no regular physical activity or exercise. Individuals with SCI are nearly 1.5 times more likely to lead sedentary lives than the general population and demonstrate significantly lower physical activity levels compared to individuals with other chronic diseases.10 Critically, everyday activities are not enough to maintain cardiovascular fitness in people with SCI, necessitating targeted exercise interventions. This "physical activity participation gap" presents a significant health crisis for individuals living with SCI and can initiate and exacerbate secondary conditions while dampening psychological well-being and quality of life (QoL). Exercise is an effective non-pharmacologic intervention to improve cardiometabolic risk factors, reduce risk for chronic and secondary conditions, and enhance psychosocial well-being. However, various barriers, such as accessibility, transportation, costs, and motivation, hinder exercise participation for those with SCI, underscoring the urgent need to provide better access to exercise experiences for this population.

Virtual reality (VR) gaming has become increasingly integrated into interventions targeting physical, neurocognitive, and psychological conditions, concurrently addressing issues like access, cost, and motivation. VR-mediated exercise interventions report strong adherence, reduced perception of effort and fatigue, and increased enjoyment of exercise participation. A global survey by the American College of Sports Medicine concluded that remote, home-based exercise, including virtual exercise, is the top fitness trend following the COVID-19 pandemic. However, while the likely benefit of home-based virtual exercise platforms for mobility impaired users is acknowledged all interventions to date have employed systems designed for able-bodied individuals. Remarkably, there has yet to be a virtual exercise platform specifically informed by input from, and exercise needs of, individuals with SCI. Further, while laboratory studies have established the potency of virtual exercise for individuals with SCI, there has yet to be a prospective study of the feasibility or cardiometabolic efficacy of a home-based virtual exercise intervention in this population. The current study assembles expertise in SCI physical health, home-based virtual reality intervention, and Lived Experience to address the abovementioned gaps by examining the feasibility and prospective efficacy of the low-cost, immersive, interactive VR exercise platform - VR-Move, deployable for self-directed use within individual homes. The project team has substantial experience and strong preliminary data supporting development and deployment of home-based immersive VR physical activity interventions for individuals with SCI. Study design is supported by a user-centered development approach (community-based participatory research) preliminary data, and a home-based technology paradigm successfully implemented by the current research team in multiple ongoing longitudinal studies with persons with SCI. The proposed study represents an important, sustainable step in promoting cardiometabolic health among people with SCI.

This proposal has integrated design elements suggested during the previous review cycle; centrally, the investigators have modified our clinical trial design with direct input from our biostatistical team to be a crossover design with a 4-week baseline control phase followed by a longer intervention phase of 12-weeks. The investigators will obtain repeated measurements at baseline (0-week), pre-intervention (4-weeks), mid-intervention (10-weeks), and post-intervention (16-weeks) which are indeed critical to understanding the longer-term impact of the intervention. The investigators have also clarified VR refinement procedures and the place of the current intervention in the larger VR pain-intervention literature. The investigators believe that these and other changes, as well as our new exciting preliminary findings, further serve to demonstrate that this novel platform has potential to meaningfully impact the health and quality of life in individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* be low risk for developing a cardiovascular event during vigorous exercise according to ACSM
* be at least 18 years of age;•
* ASIA level A-D;
* wheelchair use for at least 75% of community mobility (non-ambulatory);
* report low amounts of physical activity as determined by the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD). Participants whose combined scores for item 3 (moderate sport or recreation) and 4 (strenuous sport or recreation) ≤10 MET hours per week, will be considered physically inactive.

Exclusion Criteria:

* consistent or activity-exacerbated upper extremity pain of at least 4/10;
* angina or myocardial infarction within the last year, or other major barriers to upper-extremity exercise;
* inability to elevate arms above 45°,
* significant spasticity
* complete upper extremity impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
aerobic capacity | Enrollment to the end of the 12 week-intervention (16 weeks total)
  Participants will perform a Price and Campbell upper body ergometer test, to estimate cardiorespiratory exercise capacity. The Price and Campbell upper body ergometer test is a multistage cardiorespiratory measure that begins with an initial 2-minute warm-up period of zero-Watt (W) resistance on an upper body ergometer. Following the initial warm-up period, 30 W of resistance will be applied at a crank rate of 60 rpm for 2 minutes, representing stage one of the test. All subsequent stages are progressed incrementally in 30 W intervals at 60 rpm at 2-minute intervals until volitional exhaustion. Peak cardiorespiratory capacity (VO2peak) will be measured in ml/kg body weight.
Brief Pain Inventory | Week 10 and week 16
  The Brief Pain Inventory - Short Form (BPI-sf) is a 9-item self-administered questionnaire used to evaluate the domains of severity and pain interference. Worst, least, average, and current pain intensity and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10-point scale. A 2-point change in worst pain is considered clinically relevant.
Patient Health Questionnaire-9 (PHQ-9) | Week 10 and week 16
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The nine items are rated based on frequency of occurrence in the past two weeks "not at all" (0) to "everyday" (3) and summed. Total scores of 5, 10, 15, and 20 represent cut-points for mild, moderate, moderately severe and severe depression, respectively.
• Treatment Evaluation Inventory-short form (TEI) | End of intervention (Week 16)
  The TEI short form is a 9-item acceptability rating scale. Each statement is rated on a five-point Likert-type scale (1= Strongly Disagree to 5= Strongly Agree). Participants answer statements regarding how reasonable the intervention will be, how likely they would implement the intervention, and how effective they believed the intervention to be
Usefulness, Satisfaction, and Ease of Use Questionnaire (USE) | End of intervention (Week 16)
  The USE measures the subjective usability of a product or service. It is a 30-item survey that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. The USE questionnaire uses 27 questions with the Likert scale (1 = strongly disagree to 7 - strongly agree), with users answering questions split into 4 domains: Usefulness (8 items, score 8-56), Ease of Use (11 items, score 11-77), Ease of Learning (4 items, score 4-27) and Satisfaction (7 items, score 7-49). Item scores will be converted to a 0-100 scale with domains averaged for a total "utility" score. The positive limit of acceptable usability of the system will be defined as 50.
Simulator Sickness Questionnaire (SSQ) | End of intervention (Week 16)
  The most common reported measure of cybersickness symptoms is the Simulator Sickness Questionnaire (SSQ). The SSQ was developed to measure sickness in the context of simulation and was derived from a measure of motion sickness. Sixteen items scored 0 (none) to 3 (severe) are totaled for an overall sickness rating. Symptom severity are classified by scores such that <5 = negligible symptoms, 5-10 = minimal symptoms, 10-15 = significant symptoms with 15-20 symptoms of concern and >20 a "bad intervention.
Numeric rating scale (NRS_Pain) Pain | From beginning of intervention (week 4) through end of intervention (week 16)
  Participants will rate pain, on a 0-10 Likert scale (0 = none; 10=extreme) at beginning and end of each VR engagement (captured within the system with real-time communication to study team). Within session changes in pain, mood and nausea will be obtained during the trial. A change in pain of >30% from baseline or 2-point decrement in mood/increase in nausea will facilitate team contact and consultation with the study physician, as needed.
Numeric Rating Scale (NRS-Mood) | From beginning of intervention (week 4) through end of intervention (week 16)
  Participants will rate mood , on a 0-10 Likert scale (0 = none; 10=extreme) at beginning and end of each VR engagement (captured within the system with real-time communication to study team). Within session changes in pain, mood and nausea will be obtained during the trial. A change in pain of >30% from baseline or 2-point decrement in mood/increase in nausea will facilitate team contact and consultation with the study physician, as needed.
Numeric Rating Scale Nausea (NRS_Neausea) | From beginning of intervention (week 4) through end of intervention (week 16)
  Participants will rate nausea, on a 0-10 Likert scale (0 = none; 10=extreme) at beginning and end of each VR engagement (captured within the system with real-time communication to study team). Within session changes in pain, mood and nausea will be obtained during the trial. A change in pain of >30% from baseline or 2-point decrement in mood/increase in nausea will facilitate team contact and consultation with the study physician, as needed.

SECONDARY OUTCOMES:
Blood Pressure | Enrollment, 4 weeks, 12 weeks and 16 weeks
  Resting systolic and diastolic pressure will be measured with an Omron automated blood pressure monitor (Model BP786, Omron Healthcare, Inc., Miami, FL).
Central Adiposity | Enrollment, 4 weeks, 12 weeks and 16 weeks
  Waist and hip circumference will be measured with a Gulick tape measure (Model 67020, FitnessMart, Gays Mills, WI)-reported in cm.
Fasting blood glucose | Enrollment, 4 weeks, 12 weeks and 16 weeks
  Fasting blood glucose will be measured with an Abbott Cholestech LDX Finger stick System (Abbott, Chicago, IL). Only certified personnel will perform the finger stick procedures. Because the nature of the physical blood specimens to be collected for the proposed project are routine point of care finger sticks, we will not need to store the blood data for longer than seven (7) to ten (10) minutes. Immediately after the finger stick is collected, the blood will be placed into the Alere Cholestech LDX analyzer, which will then analyze and provide the blood glucose values for the participant within the 10-min timeframe.
Fasting blood lipid profiles | Enrollment, 4 weeks, 12 weeks and 16 weeks
  Fasting blood lipid profiles will be measured with an Abbott Cholestech LDX Finger stick System (Abbott, Chicago, IL). Because the nature of the physical blood specimens to be collected for the proposed project are routine point of care finger sticks, we will not need to store the blood data for longer than seven (7) to ten (10) minutes. Immediately after the finger stick is collected, the blood will be placed into the Alere Cholestech LDX analyzer, which will then analyze and provide the lipid values for the participant within the 10-min timeframe.

OTHER OUTCOMES:
Exercise Self Efficacy Scale (ESE) | Enrollment, 4 weeks, 12 weeks and 16 weeks
  This self-report measures the construct of self-efficacy, or personal beliefs in one's capabilities relating to exercise participation in individuals with SCI. The 10 items are rated from 1 = "not at all" to 4- Exactly true" and items are summed for a total score. Self-efficacy is cited as the most critical personal factor to behavior change.
SCI Quality of Life Resilience, SCIQoL_RES | Enrollment, 4 weeks, 12 weeks and 16 weeks
  The Resilience short form bank contains 8 items that address issues such as motivation, coping, and acceptance. Scores are converted to T-scores
SCI Quality of Life Positive Affect and Well-being, PAWB | Enrollment, 4 weeks, 12 weeks and 16 weeks
  The 10-item bank addresses aspects of a person's life that relate to a sense of well-being, life satisfaction, or an overall sense of purpose and meaning.
  Scores are converted to T-scores
SCI Quality of Life pain interference; SCIQoL_PI | Enrollment, 4 weeks, 12 weeks and 16 weeks
  The SCI-QoL Pain Interference short form (10 items) is versions of the PROMIS Pain Interference item banks, that have been optimized for individuals with SCI.
  Scores are converted to T-scores
Satisfaction with Life Scale (SWLS) | Enrollment, 4 weeks, 12 weeks and 16 weeks
  The SWLS is a 5 item, 7-point Likert response scale. The possible range of scores is 5-35, with a score of 20 representing a neutral point on the scale.
General Sleep Disturbance Scale, GSDS | Enrollment, 4 weeks, 12 weeks and 16 weeks
  The GSDS is a 21-item scale was designed to evaluate the incidence and nature of sleep disturbances. The GSDS queries respondents regarding the frequency with which they've experienced certain sleep difficulties within the previous week. Respondents use an eight-point, Likert-type scale ranging from 0 (meaning "never") to 7 ("every day") to respond to each item. The total score for the scale ranges between 0 and 147, with higher scores indicating a higher frequency of sleep disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University Health Science Building, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the FAIR practices and standards for sharing of SCI data, we will share final individual participant outcomes and metadata organized as recommended by ODC-SCI, using formatting standards established by the ODC-SCI. By following these recommendations, we will ensure that our data may be harmonized with other clinical studies and has passed community quality checks. All experimental data will be accompanied by a detailed experimental protocol and additional data and metadata. The protocols will be linked to the experimental data both in the publication and the data sharing platform. ODC-SCI requires the publication of a data dictionary that defines all variables present in the data set in a standard format.
Supporting Information: Study Protocol, SAP